CLINICAL TRIAL: NCT05721742
Title: Evaluating the Impact of Including Virtual Dietary Education Within an Electronic Irritable Bowel Syndrome Pathway
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Research Nova Scotia (Unknown)
Responsible Party: Principal Investigator, Jennifer Jones, Gastroenterologist, Associate Professor, Department of Medicine, Dalhousie University, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 53363
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pre-existing online group education program for IBS (Active Comparator): This arm will be enrolled in the online course run by Happy Bellies Nutrition https://www.happybelliesnutrition.com/ibs-gentle-group-program. The Happy Bellies nutrition course has 5.5 hours of total video content and optional biweekly group calls via Zoom (45-minutes per session). This course is designed to take 12 weeks to complete. The participants would have access to the content for one year.
  Interventions: Other: IBS Group Online Session
- virtual dietitian consults for IBS patients (Experimental): This arm will receive consults with a virtual dietitian (60 minutes initial + 4 x30-minute follow-up appointment) by a dietitian who has had additional training in the dietary management of IBS.
  Interventions: Other: virtually administered dietitian consults for IBS patients.

INTERVENTIONS:
Other: virtually administered dietitian consults for IBS patients. — Participants will receive virtual one on one consults with a dietitian who has training in the dietary management of IBS.
  Arms: virtual dietitian consults for IBS patients
Other: IBS Group Online Session — IBS online group session run by Happy Bellies Nutrition
  Arms: pre-existing online group education program for IBS

SUMMARY:
Irritable bowel syndrome is a functional bowel disorder that affects many Canadians. The syndrome involves abdominal pain and change in frequency or form of bowel movements, and these symptoms can lead to a decreased quality of life for patients. Primary care physicians are dissatisfied with current referral processes, and patients may wait a long time to receive the correct diagnosis. Diet is known to exacerbate symptoms of IBS. In Canada, accessing dietary treatment for IBS is a challenge due to lack of resources. Some patients lack access to dietary interventions, and others are given advice that is not evidenced based. Use of eHealth technology, such as virtual education delivered by a dietician, may allow for more widespread access to dietary interventions for IBS. Virtual education can include one on one dietary education, online group-based education, and the use of apps. Currently, there is a gap in knowledge whether dietary intervention for IBS, delivered virtually by a dietician, is effective in treating IBS.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent abdominal pain on average at least 1 day/ week in the last 3 months associated with two or more of the following criteria: related to defecation, or association with a change in frequency of stool or associated with a change in form (appearance) of stool
* Willingness to change diet
* Access to a device for accessing virtual dietary education

Exclusion Criteria:

* New onset symptoms within past year in age 50 and above
* Rectal bleeding
* Inflammatory Bowel Disease
* Unexplained recent weight loss
* Gastrointestinal surgery with removal of gallbladder or segments of the bowel
* Having an eating disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
IBS Symptom Severity | Baseline
  IBS Symptom Severity as measured by the "IBS Symptom Severity Score". Minimum: 75, Maximum: >300. Mild, moderate and severe cases are indicated by scores of 75 to 175, 175 to 300 and > 300 respectively.
IBS Symptom Severity | 5 months post-randomization
  IBS Symptom Severity as measured by the "IBS Symptom Severity Score". Minimum: 75, Maximum: >300. Mild, moderate and severe cases are indicated by scores of 75 to 175, 175 to 300 and > 300 respectively.
IBS Specific Quality of Life | Baseline
  IBS Specific Quality of Life as measured by the "IBS Quality of Life Questionnaire". Minimum: 0, Maximum: 100. Higher scores indicating better IBS specific quality of life.
IBS Specific Quality of Life | 5 months post-randomization
  IBS Specific Quality of Life as measured by the "IBS Quality of Life Questionnaire". Minimum: 0, Maximum: 100. Higher scores indicating better IBS specific quality of life.
Patient Quality of Life | Baseline
  Patient Quality of Life as measured by the "EQ 5D 5L Questionnaire". This questionnaire comprises the following five dimensions (ie. five questions): mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension (question) has 5 levels (possible answers): 1-no problems, 2-slight problems, 3-moderate problems, 4-severe problems and 5-extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement. This results in a 1-digit number that expresses the level selected for that dimension, and the digits for the five dimensions are combined into a 5-digit number that describes the patient's health state. There is also a visual analog scale which asks the patient to rate their overall health from 0-100, with 0 being the worst, and 100 being best possible health.
Patient Quality of Life | 5 months post-randomization
  Patient Quality of Life as measured by the "EQ 5D 5L Questionnaire". This questionnaire comprises the following five dimensions (ie. five questions): mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension (question) has 5 levels (possible answers): 1-no problems, 2-slight problems, 3-moderate problems, 4-severe problems and 5-extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement. This results in a 1-digit number that expresses the level selected for that dimension, and the digits for the five dimensions are combined into a 5-digit number that describes the patient's health state. There is also a visual analog scale which asks the patient to rate their overall health from 0-100, with 0 being the worst, and 100 being best possible health.
Total number Inpatient services in the last 3 months | Baseline
  Total number of inpatient services (admissions) in the last 3 months the patient has received, using an adaptation of the Client Services Receipt Inventory (CSRI). The PI will create a questionnaire containing the Service Receipt (Section 4) questions of the CSRI.
Total number Inpatient services in the last 3 months | 5 months post randomization
  Total number of inpatient services (admissions) in the last 3 months the patient has received, using an adaptation of the Client Services Receipt Inventory (CSRI). The PI will create a questionnaire containing the Service Receipt (Section 4) questions of the CSRI.
Total number Outpatient appointments in the last 3 months | baseline
  Total number of outpatient services (outpatient appointments) in the last 3 months the patient has received, using an adaptation of the Client Services Receipt Inventory (CSRI). The PI will create a questionnaire containing the Service Receipt (Section 4) questions of the CSRI.
Total number Outpatient appointments in the last 3 months | 5 months post randomization
  Total number of outpatient services (outpatient appointments) in the last 3 months the patient has received, using an adaptation of the Client Services Receipt Inventory (CSRI). The PI will create a questionnaire containing the Service Receipt (Section 4) questions of the CSRI.
Volume of referrals to Dietician | 5 months post-randomization
  Volume of referrals sent to the Virtual Dietician led 1 on 1 education session
Volume of referrals to Online Group Session | 5 months post-randomization
  Volume of referrals sent to the online IBS group session, run by Happy Bellies Nutrition
Patient satisfaction with the Virtual Dietician led 1 on 1 education session | 5 weeks post-randomization
  Patient satisfaction with the Virtual Dietician led 1 on 1 education session measured via questionnaires that were written by the study PI. The following statements will be presented, answers will follow a 5-point Likert scale where 1-strongly disagree 2-disagree 3-neutral 4-agree 5-strongly agree:
  1. I feel confident managing my IBS
  2. Overall, I was satisfied receiving dietary education through telehealth
  3. It was easy to ask questions and get answers
  4. I felt comfortable communicating with the dietitian using the telehealth system
  5. It was easy to use the technology to access the services
  6. I had no concerns about the privacy of my personal data
  7. I would recommend this service to friends and family
Volume of 1 on 1 dietary consults completed | 5 months post-randomization
  Volume of 1 on 1 dietary consults completed, records kept by study dieticians
Number of online modules competed for Online Group Session | 5 months post-randomization
  Number of online modules competed for Online Group Session
Number of sessions compared to proposed | 5 months post-randomization
  Number of virtual dietician led 1 on 1 education sessions compared to proposed
Number of Modules accessed | 5 months post-randomization
  Number of Modules accessed for Online group session program run by Happy Bellies Nutrition
Number of Modules completed | 5 months post-randomization
  Number of Modules completed for Online group session program run by Happy Bellies Nutrition
Percentage participation in group session | 5 months post-randomization
  Percentage of participation for Online group session program run by Happy Bellies, Nutrition measured by how many participants contributed
Quality Adjusted Life Years | 5 months post-randomization
  Quality adjusted life years as measured using the EQ 5D and client service receipt inventory

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, N.S., Canada

IPD SHARING:
Plan to Share IPD: No